CLINICAL TRIAL: NCT02432014
Title: DCISR for Adaptive Intervention Models in Children's Mental Health
Brief Title: Parent Preferences and Family Engagement in a Conduct Problems Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Michigan Department of Community Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1006S83774; P20MH085987 (NIH)
Record Dates: First submitted 2015-04-03; First posted 2015-05-01 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Conduct Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PMTO-PTC Group clinic-based (Other): PMTO-PTC = Oregon Parent Management Training program, Parenting Through Change groups provided at a clinic.
  Interventions: Behavioral: PMTO-PTC Group clinic-based
- PMTO Individual home-based (Other): PMTO = Oregon Parent Management Training program, delivered individually in the home.
  Interventions: Behavioral: PMTO Individual home-based
- PMTO Individual clinic-based (Other): PMTO = Oregon Parent Management Training program, delivered individually at a clinic.
  Interventions: Behavioral: PMTO Individual clinic-based
- Services as Usual (Other): Usual child-centered services (i.e. therapy) provided by the agencies at a clinic.
  Interventions: Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: PMTO-PTC Group clinic-based
  Other Names: PMTO-Parenting Through Change - Group
  Arms: PMTO-PTC Group clinic-based
Behavioral: PMTO Individual home-based
  Other Names: Oregon Parenting Management Training - Individual @ home
  Arms: PMTO Individual home-based
Behavioral: PMTO Individual clinic-based
  Other Names: Oregon Parent Management Training - Individual @ clinic
  Arms: PMTO Individual clinic-based
Behavioral: Services as Usual
  Arms: Services as Usual

SUMMARY:
The purpose of this study is to gain a better understanding of family preferences for and engagement in services.

DETAILED DESCRIPTION:
The overarching goal of this pilot project is to elucidate factors that influence families' engagement in indicated prevention/early intervention programming for youth conduct problems. We will explore factors previously shown to influence engagement, including parent motivational cognitions, family context variables, and preferences for intervention type. Study aims are organized around a randomized preference trial with a parallel hybrid design structure (see Abikoff, 2001). Families with youth ages 5-12, referred to community mental health clinics in Michigan, will be invited to participate in a prevention study. Families who chose to participate were assigned at random to preference (i.e. choice) or no preference (i.e. no choice) conditions. Those randomly assigned to the preference condition were allowed to choose between four intervention options: clinic-based services-as-usual (youth intervention); individual, home-based Oregon Parent Management Training (PMTO; Patterson, 2005), individual, clinic-based PMTO, and in-person group-based PMTO (Parenting Through Change; Forgatch & DeGarmo, 1999). Families in the no-choice condition were randomly assigned to one of the same four conditions.

ELIGIBILITY:
Inclusion Criteria:

* Families with at least one child between the ages of 5 and 12.
* Referral to community mental health clinic (specifically, to one of the project partner clinics)

Exclusion Criteria:

* Active psychosis
* Serious child mental health diagnosis
* Open child protection case for abuse or neglect

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Family Interaction Task (FIT) | 1 year
  Parent(s) and child participate in a number of activities which are observed and coded based on parent-child interactions.
Strengths and Difficulties Questionnaire | 1 year
  Parent and Teacher Report
Brief Symptom Inventory 18 (BSI-18) Questionnaire | 1 year
  Parent Report
Perceptions of Intervention Benefits and Barriers Questionnaire | 1 year
  Parent Report
Parent Locus of Control Questionnaire | 1 year
  Parent Report
Perceived Susceptibility & Severity Questionnaire | 1 year
  Parent Report
Perceived Need to Improve Parenting Questionnaire | 1 year
  Parent Report
Child Service Utilization Summary Questionnaire | 1 year
  Parent Report

CONTACTS AND LOCATIONS:
Overall Officials: Gerald August, Ph.D., Principal Investigator — University of Minnesota - P20-Center Director (PI); Abigail Gewirtz, Ph.D., Principal Investigator — University of Minnesota - Pilot Project PI
Locations (1):
- Center for Personalized Prevention Research in Children's Mental Health, Minneapolis, Minnesota, United States